CLINICAL TRIAL: NCT01408979
Title: Postpartum Prophylaxis With Short Course Magnesium Sulfate in Severe Preeclampsia: a Randomized Clinical Trial
Brief Title: Effectiveness Study of Short Course of Magnesium Sulfate for Severe Preeclamsia
Acronym: MgSO4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Principal Investigator, Leila Katz, Obstetrical ICU obstetrical coordinator; MD , PhD, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MgSO4
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-04

CONDITIONS: Severe Preeclampsia
Keywords: Severe preeclampsia; magnesium sulfate; anticonvulsivant
MeSH Terms: conditions — Pre-Eclampsia | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 12 hours of magnesium sulfate (Experimental): Patients in this group will have magnesium sulfate administered for 12 hours after delivery
  Interventions: Drug: Magnesium sulfate 12 hours
- 24 hours of magnesium sulfate (Active Comparator): Patients in this group will have magnesium sulfate administered for 24 hours after delivery
  Interventions: Drug: Magnesium sulfate 24 hours

INTERVENTIONS:
Drug: Magnesium sulfate 12 hours — Magnesium sulfate, 1g/h, (10% solution), for 12 hours
  Arms: 12 hours of magnesium sulfate
Drug: Magnesium sulfate 24 hours — Magnesium sulfate, 1g/h, (10% solution), for 24 hours
  Arms: 24 hours of magnesium sulfate

SUMMARY:
Magnesium sulfate is the ideal drug for seizures prophilaxis in preeclampsia. The ideal duration of this treatment after delivery is still to be established. The hypothesis is that in stable patients a shorter course of treatment is possible without prejudice to the mother.

DETAILED DESCRIPTION:
Magnesium sulfate (MgSO4) is certainly the ideal drug for prevention and control of eclamptic seizures. However, there is no consensus on the appropriate duration of prophylaxis with this anticonvulsant postpartum.The objective of the present study is to compare effectiveness of 12 hours of magnesium sulfate versus 24 hours (standard treatment) in stable patients with preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Pre-eclampsia;
* Puerperium.

Exclusion Criteria:

* Associated maternal diseases;
* Use of illicit drugs or other medications that might interfere with maternal hemodynamics;
* Contraindications to the use of magnesium sulfate: drug hypersensitivity, oliguria with urine output below 25ml/h; anuria (absent urine output), myasthenia gravis.

Ages: 11 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Need to continue therapy for another 12 hours. | 24 hours
  Defined as the need to continue therapy for another 12 hours, this will occur when after the first 12 hours of magnesium sulfate therapy the patient has severe hypertension, unsatisfactory diureses or has signs or symptoms of iminent eclampsia.

SECONDARY OUTCOMES:
Satisfaction | 24 hours
  Patients satisfaction with the duration of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Melania M Amorim, MD; PhD, Principal Investigator — IMIP
Locations (1):
- IMIP, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Diaz V, Long Q, Oladapo OT. Alternative magnesium sulphate regimens for women with pre-eclampsia and eclampsia. Cochrane Database Syst Rev. 2023 Oct 10;10(10):CD007388. doi: 10.1002/14651858.CD007388.pub3. PMID 37815037
- [Derived] Maia SB, Katz L, Neto CN, Caiado BV, Azevedo AP, Amorim MM. Abbreviated (12-hour) versus traditional (24-hour) postpartum magnesium sulfate therapy in severe pre-eclampsia. Int J Gynaecol Obstet. 2014 Sep;126(3):260-4. doi: 10.1016/j.ijgo.2014.03.024. Epub 2014 May 10. PMID 24890747